CLINICAL TRIAL: NCT05116215
Title: To Evaluate the Safety of Treating Autoimmune Diseases With Molecular Hydrogen Supplement
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HoHo Biotech (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-B202105106
Record Dates: First submitted 2021-10-08; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Hydrogen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydrogen inhalation (Experimental): Participants in the gas group will then undergo exposure to 2% H2 in medical air via a high flow nasal cannula for either 1 (n=3), 2 (n=3) or 4 (n=3) hours every day for one month.
  Interventions: Drug: Hydrogen
- Hydrogen capsules (Experimental): Participants in capsule group will receive either 1 (n=3), 3 (n=3) or 6 (n=3) capsules every day for one month.
  Interventions: Drug: Hydrogen
- Hydrogen water (Experimental): Participants in the water group will be suggested to drink 1 L hydrogen-rich water every day for one month.
  Interventions: Drug: Hydrogen

INTERVENTIONS:
Drug: Hydrogen — Hydrogen supplement

SUMMARY:
The supplementation of hydrogen molecules as an aid, adjuvant, may speed up recovering the course of the disease. The purpose of this study is to determine the safety and possible efficacy of hydrogen supplements in different formula and dose exposures for a clinical study in rheumatologic patients. Patients will receive a different dosage of either hydrogen capsules, hydrogen gas or hydrogen-rich water with their conventional treatment for a month. Investigators will test for any changes in haematologic, urine analysis and health status during and following the exposure period.

DETAILED DESCRIPTION:
Hydrogen supplement has been shown to have significant removing effects on free radicals. International clinical trials have shown promise that hydrogen molecules may reduce chronic inflammatory and then speed up recovering the course of the disease.

The purpose of this study is to determine the safety and possible efficacy of hydrogen supplements in different formula and dose exposures for a clinical study in rheumatologic patients.

Study design: 27 rheumatologic patients will be recruited from the Tri-Service General Hospital for this study. Participants will be screened by doctors for their eligibility and undergo a series of tests (questionnaires and examinations). Consenting participants will then be allocated into 3 groups by different dosage forms (Gas, n=9; Water, n=9; Capsules, n=9). Participants in the gas group will then undergo exposure to 2% H2 in medical air via a high flow nasal cannula for either 1 (n=3), 2 (n=3) or 4 (n=3) hours every day for one month. Participants in capsule group will receive 1 (n=3), 3 (n=3) or 6 (n=3) capsules every day for one month. Participants in the water group will be suggested to drink 1 L hydrogen-rich water every day for one month. Participants will be examined their regular haematology, urine and health status before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80
* Able to compliant with the protocol
* Able to return to the hospital regularly

Exclusion Criteria:

* Pregnancy
* Expected pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-08-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Routine | Change from Baseline Blood Routine at Day 28
  Numerical change in Blood Routine
Change in Urine Routine | Change from Baseline Urine Routine at Day 28
  Numerical change in Urine Routine
Health Assessment Questionnaire Disability Index, HAQ-DI | Change from Baseline HAQ-DI at Day 28
  Questionnaire
Disease Activity Score, DAS 28 | Change from Baseline DAS 28 at Day 28
  A score of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No